CLINICAL TRIAL: NCT06947902
Title: Optimizing High Flow Nasal Cannula Oxygenation in Pediatric Airway Procedures: a Randomized Study
Brief Title: Optimizing High Flow Nasal Cannula Oxygenation in Pediatric Airway Procedures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Zhen Huang, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC-MS-25-0028
Record Dates: First submitted 2025-04-17; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Airway Disorder
Keywords: High Flow Nasal Cannula (HFNC)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- High flow (Experimental)
  Interventions: Device: High flow
- Low Flow (Experimental)
  Interventions: Device: Low Flow

INTERVENTIONS:
Device: High flow — The High Flow Nasal Cannula (HFNC) device (Vapotherm) will be placed through the nostrils for oxygen (2L/kg per min with max of 45L)
  Arms: High flow
Device: Low Flow — The High Flow Nasal Cannula (HFNC) device (Vapotherm) will be placed through the nostrils for oxygen (0.5L/kg per min with max of 5L)
  Arms: Low Flow

SUMMARY:
The purpose of this study is to investigate which flow rate (higher versus lower) is most effective at increasing apneic time and preventing greater than 5% drop in desaturation, as well as assessing transcutaneous carbon dioxide (CO2) levels during airway procedures in children

ELIGIBILITY:
Inclusion Criteria:

* undergoing laryngoscopy and bronchoscopy procedures at Children's Memorial Hermann Hospital (CMHH)
* weight greater than or equal to 5 kilograms and using flow rates between 5 to 45 liters per minute (BTPS)

Exclusion Criteria:

* Emergency type cases, tracheostomy patients, unrepaired cyanotic heart disease, nasal deformity/choanal atresia, or cautery/laser type procedures

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants that show an incidence of oxygen desaturation >5 % | from start of procedure to end of procedure (about 1 hour)

SECONDARY OUTCOMES:
Apnea time measured in seconds or minutes | from start of procedure to end of procedure (about 1 hour)
Number of Participants With Surgical Interruptions Due to Desaturation | from start of procedure to end of procedure (about 1 hour)
  Number of surgical interruptions due to desaturation defined by a pause in surgical procedures due to need to provide airway intervention to improve patient's oxygen saturation, normalized to case length. Airway interventions may include LMA, bag mask ventilation, and/or endotracheal intubations
Oxygen nadir level | from start of procedure to end of procedure (about 1 hour)
Transcutaneous CO2 measurements throughout procedure | from start of procedure to end of procedure (about 1 hour)
Adverse events related to device itself (nasal pain, skin irritation) | from baseline to end of study (1 month after baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Huang, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No